CLINICAL TRIAL: NCT00830128
Title: An Open-Label Extension Safety And Efficacy Study Of Pregabalin (CI-1008) For The Treatment Of Fibromyalgia
Brief Title: A Long-Term Study To Evaluate Safety And Efficacy Of Pregabalin In Patients With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0081209
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Results first posted 2012-02-14 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2012-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pregabalin (Lyrica) (Experimental)
  Interventions: Drug: pregabalin (Lyrica)

INTERVENTIONS:
Drug: pregabalin (Lyrica) — Dosage: 300-450 mg/day (150-225 mg twice daily), oral administration, Treatment duration: 52 weeks

SUMMARY:
This study will assess the safety and efficacy of the long-term use of pregabalin at doses up to 450 mg/day in patients with fibromyalgia who have completed 16 weeks of dosing in Study A0081208 (NCT00830167).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met the inclusion criteria for the preceding fibromyalgia Protocol A0081208, and must have received pregabalin/placebo under double-blind conditions.

Exclusion Criteria:

* Patients may not participate in the study if they experienced a serious adverse event during the previous fibromyalgia Study A0081208; which was determined to be related to the study medication by the investigator or the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- Japan (19):
  - Pfizer Investigational Site, Yotukaidou, Chiba
  - Pfizer Investigational Site, Matuyama-si, Ehime
  - Pfizer Investigational Site, Iiduka, Fukuoka
  - Pfizer Investigational Site, Kobe, Hyōgo
  - Pfizer Investigational Site, Mito, Ibaraki
  - Pfizer Investigational Site, Morioka, Iwate
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Tsu, Mie-ken
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Hiki-gun, Saitama
  - Pfizer Investigational Site, Saitama-shi, Saitama
  - Pfizer Investigational Site, Shimotsuga-gun, Tochigi
  - Pfizer Investigational Site, Chiyoda-ku, Tokyo
  - Pfizer Investigational Site, Itabashi-Ku, Tokyo
  - Pfizer Investigational Site, Shinagawa-ku, Tokyo
  - Pfizer Investigational Site, Nagano
  - Pfizer Investigational Site, Osaka
  - Pfizer Investigational Site, Ōita
  - Pfizer Investigational Site, Yokohama

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081209&StudyName=A%20Long-Term%20Study%20To%20Evaluate%20Safety%20And%20Efficacy%20Of%20Pregabalin%20In%20Patients%20With%20Fibromyalgia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received the study drug in the precedent study A0081208 (NCT00830167).
Groups:
- Pregabalin: Pregabalin treatment was started at 150 mg/day in Week 0 and escalated to 300 mg/day at Week 1. After that, participants could receive a maximum dose of 450 mg/day (225 mg, twice daily) for 52 weeks. During the term of the study, the dosage was to be adjusted (dose escalation/decrease), taking safety and efficacy with respect to pain into account.
Period: Overall Study
Arm/Group | Pregabalin
Started | 106
Completed | 87
Not Completed | 19
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 7
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 2
Not completed — Family obligation | 1
Not completed — Relocation | 1
Not completed — Work obligation | 1
Not completed — Operating a vehicle | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Age, Customized [Number; unit: Participants]
  <18 years | 0
  Between 18 and 44 years | 47
  Between 45 and 64 years | 49
  >= 65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Any untoward medical occurrence in a participant who received study drug was considered an adverse event (AE), without regard to possibility of causal relationship. Treatment-emergent adverse events: those which occurred or worsened after baseline. An AE resulting in any of the following outcomes, was considered to be a serious adverse event: death; lifethreatening; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect.
Time Frame: Up to 53 weeks
Population: All participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Participants
  All-causality adverse events (AEs) | 102
  All-causality SAEs | 3

2. Secondary Outcome: Change From Baseline in Pain Visual Analog Scale (Pain VAS) Score at Endpoint
Description: The pain VAS is a horizontal line; 100 mm in length, self-administered by the patient to rate pain from 0 (no pain) to 100 (worst possible pain). The score indicates the pain intensity during the past 1 week before a visit.
  Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 52 or Study Discontinuation
Population: All participants who have taken at least 1 dose of the study medication, regardless of compliance with the study medication, and have at least 1 postbaseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
mm | -13.1 (25.3)

3. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale - Sleep Disturbance at Endpoint
Description: MOS: patient rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Sleep Disturbance subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score means greater sleep disturbance.
  Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 52 or Study Discontinuation
Population: All participants who received at least 1 dose of the study medication, regardless of compliance with the study medication, and had at least 1 postbaseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Units on a scale | -9.6 (23.3)

4. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale - Snoring at Endpoint
Description: MOS: patient rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Snoring subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score means worse symptoms.
  Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 52 or Study Discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Units on a scale | 1.9 (22.3)

5. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale - Awaken Short of Breath or With a Headache at Endpoint
Description: MOS: patient rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Awaken Short of Breath or With a Headache subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score means worse symptoms.
  Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 52 or Study Discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Units on a scale | -3.0 (23.1)

6. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale - Sleep Adequacy at Endpoint
Description: MOS: patient rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Sleep Adequacy subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score means greater sleep adequacy.
  Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 52 or Study Discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Units on a scale | 4.2 (21.3)

7. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale - Quantity of Sleep at Endpoint
Description: MOS: patient rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Quantity of Sleep subscales rated 0 to 24 (number of hours slept). A higher score means greater quantity of sleep.
  Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 52 or Study Discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
hours | 0.3 (1.2)

8. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale - Somnolence at Endpoint
Description: MOS: patient rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Somnolence subscales rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score means worse symptoms.
  Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 52 or Study Discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Units on a scale | 7.2 (24.0)

9. Secondary Outcome: Change From Baseline in Medical Outcomes Study (MOS) Sleep Scale - Overall Sleep Problems Index at Endpoint
Description: MOS: patient rated questionnaire to assess sleep quality and quantity. Consists of 9-item overall sleep problems index (length of time to fall asleep, how many hours of sleep each night during past 4 weeks); The MOS Overall Sleep Problems Index rated 1 (all the time) to 6 (none of the time). Scores are transformed (actual raw score minus lowest possible score) divided by possible raw score range multiplied by 100; total score range = 0 to 100. A higher score means worse symptoms.
  Change = mean scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 52 or Study Discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Units on a scale | -3.7 (15.7)

10. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Scale - Optimal Sleep at Endpoint
Description: MOS-Sleep is a patient-rated questionnaire to assess sleep quality and quantity. Optimal sleep component is derived from Sleep Quantity average hours of sleep each night during the past 4 weeks. Number of participants with response = YES if sleep quantity is 7 or 8 hours per night or response = NO if sleep quantity is < 7 hours per night.
Time Frame: Week 52 or Study Discontinuation
Population: as for outcome 3
Measure: Number; unit: Paticipants
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Paticipants
  Yes | 26
  No | 80

11. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) - Total Scores at Endpoint
Description: FIQ is a 20-item patient-reported outcome instrument designed to assess health status, progress, and outcomes in patients with fibromyalgia (10 subscales; 11 questions). Scores range from 0 to 100 with higher scores indicating more impairment.
  Change = mean FIQ scores at observation minus mean scores at baseline.
Time Frame: Baseline, Week 52 or Study Discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Units on a scale | -4.9 (17.2)

12. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) - Subscale Score at Endpoint
Description: as for outcome 11
Time Frame: Baseline, Week 52 or Study Discontinuation
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin
Number analyzed (Participants) | 106
Units on a scale
  Physical Functioning | -0.2 (2.0)
  Feel Good | -0.4 (2.7)
  Work Missed | -0.5 (2.8)
  Difficulty Working | -0.7 (2.6)
  Pain | -1.0 (2.3)
  Fatigue | -0.3 (1.9)
  Morning Tiredness | -0.6 (2.2)
  Stiffness | -0.7 (2.5)
  Anoxiouness | -0.3 (2.6)
  Depression | -0.2 (2.6)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin
Serious Adverse Events (participants affected / at risk) | 3/106
Other Adverse Events (participants affected / at risk) | 92/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=106)
Tuberculosis (Infections and infestations) | 1
Crush Injury (Injury, poisoning and procedural complications) | 1
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1
Neuropathy Peripheral (Nervous system disorders) | 1
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=106)
Abdominal pain upper (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 23
Nausea (Gastrointestinal disorders) | 7
Oedema peripheral (General disorders) | 9
Nasopharyngitis (Infections and infestations) | 33
Fall (Injury, poisoning and procedural complications) | 6
Weight increased (Investigations) | 21
Back pain (Musculoskeletal and connective tissue disorders) | 6
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 9
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 28
Headache (Nervous system disorders) | 12
Somnolence (Nervous system disorders) | 31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.